CLINICAL TRIAL: NCT00224276
Title: Prevalence and Incidence of Diabetes Mellitus Among Patients Treated With Atypical and Conventional Antipsychotics
Brief Title: Prevalence of Diabetes Mellitus Among Patients Treated With Atypical and Conventional Antipsychotics
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Other Study IDs: RIS-USA-302
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Bipolar Disorder; Diabetes Mellitus
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This pilot study hypothesizes that diagnosed and undiagnosed prevalence of diabetes mellitus may differ across antipsychotioc medications in a community mental health center. The study further hypothesizes that control of diabetes among diagnosed cases may be suboptimal.

DETAILED DESCRIPTION:
Study of longitudinal incidence proved impractical within the limitations of the project.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with antipsychotic medication at a community mental health center

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University